CLINICAL TRIAL: NCT05401552
Title: The Impact of Phosphate Bioavailability on the Hormonal Response to a Breakfast Meal in Healthy Humans
Brief Title: Phosphate Bioavailability Hormonal Response to a Breakfast Meal in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Rachel Holden, Professor, Clinical Evaluation Research Unit at Kingston General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DMED-2049-17
Record Dates: First submitted 2022-04-27; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Phosphate Overload
MeSH Terms: interventions — Meals

STUDY DESIGN:
Intervention Model Description: cross-over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convenience breakfast meal (Active Comparator): One cheese tea biscuit and Eggo waffle
  Interventions: Other: Meal
- Healthy breakfast meal (Active Comparator): One cup of All-Bran breakfast cereal with milk and a piece of fruit
  Interventions: Other: Meal

INTERVENTIONS:
Other: Meal — Comparison of two breakfast meals containing the same amount of phosphorus but one in the form of inorganic additives

SUMMARY:
Convenience food is enhanced with phosphate additives in order to modify taste and texture and for preservation. The purpose of this study is to measure the response of phosphate-related hormones to two different types of breakfast meals that contain the same amount of phosphate but in different forms. This study is a cross-over design.

DETAILED DESCRIPTION:
In the first meal, the participant will consume a standard convenience breakfast meal comprised of a cheese tea biscuit and two Eggo waffles. The amount of phosphorus contained in this meal is 700 mg and the majority of this phosphate would be in the form of phosphate additives. Urine and blood will be collected before and after consumption of the meal to measure how the body responds to the meal. Specifically, levels of phosphate, calcium, creatinine (measure of kidney function) and three hormones involved in phosphate regulation (parathyroid hormone, fibroblast growth factor-23 and vitamin D) will be measured in each blood sample. Creatinine, calcium and phosphate will be measured in each urine sample. The second meal will also contain 700 mg of phosphorus and similar caloric content but in a healthy breakfast meal that does not contain any phosphate additives, consisting of one cup of All-Bran breakfast cereal with milk and a piece of fruit. The same blood and urine tests will be assessed after the second meal.

ELIGIBILITY:
Inclusion Criteria

* healthy

Exclusion Criteria:

* kidney disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Urine phosphate excretion | 4 hours
  The amount of phosphate excreted into the urine

SECONDARY OUTCOMES:
urine calcium excretion | 4 hours
  The amount of calcium excreted into the urine
Blood phosphate and calcium | 3 hours
  blood levels of phosphate and calcium
Parathyroid hormone | 4 hours
  blood level of parathyroid hormone

CONTACTS AND LOCATIONS:
Overall Officials: Rachel M Holden, MD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Queen's University, Kingston, Ontario
  - Rachel Holden, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
undecided